CLINICAL TRIAL: NCT06794840
Title: Optimizing a Just-in-Time Adaptive Intervention to Increase Uptake of Chemsex Harm Reduction Services in MSM: A Micro-randomized Trial
Brief Title: JomCare Study - A Harm Reduction Study
Acronym: JomCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other); Yale University (Other); National Institute on Drug Abuse (NIDA) (NIH); University of Michigan (Other); University of Texas at Tyler (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 24-047-910; R01DA061661 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-01-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: HIV; Substance Abuse Disorder
Keywords: HIV; mHealth; JITAI; Chemsex
MeSH Terms: conditions — Substance-Related Disorders; Chemsex

STUDY DESIGN:
Intervention Model Description: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) that uses an EMA-based machine learning (ML) algorithm to anticipate chemsex risk and deliver appropriate chemsex-related harm reduction and HIV prevention services when the risk is detected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Information-based engagement prompts (Experimental): Information-based engagement prompts are expected to improve participants' knowledge of harm reduction needs by providing information relevant to HIV (e.g., HIV/STI risk reduction), chemsex (e.g., safer drug use, CAD overdose prevention, drug interactions), and other topics (e.g., mental health).
  Interventions: Behavioral: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) for chemsex-related harm reduction.
- Motivation-based engagement prompts (Experimental): Motivation-based engagement prompts are expected to increase the salience of participants' beliefs about the importance of their harm reduction needs.
  Interventions: Behavioral: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) for chemsex-related harm reduction.
- Behavioral skills-based engagement prompts (Experimental): Behavioral skills-based engagement prompts are expected to improve self-efficacy and the ability to engage in intervention.
  Interventions: Behavioral: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) for chemsex-related harm reduction.
- Generic engagement prompts (Active Comparator): Generic engagement prompts are included as active comparators to the theory-driven components, as they control for the potential influence of receiving any engagement prompts. Given the aim to optimize JITAI, including generic prompts provides the mechanism for distinguishing the effects of receiving any prompt from the theory-driven prompts.
  Interventions: Behavioral: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) for chemsex-related harm reduction.
- No engagement prompt (No Intervention): No engagement prompt is included as an inactive comparator. Participants will not receive any prompt when randomized to this group. Inclusion of the "no engagement prompt" will control for the potential impact of being notified of heightened risk, which could activate any pre-existing strategies to reduce or prevent risk.

INTERVENTIONS:
Behavioral: JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) for chemsex-related harm reduction. — JomCare is a smartphone-based just-in-time adaptive intervention (JITAI) that uses an EMA-based machine learning (ML) algorithm to anticipate chemsex risk and deliver appropriate chemsex-related harm reduction and HIV prevention services when the risk is detected.
  Arms: Behavioral skills-based engagement prompts; Generic engagement prompts; Information-based engagement prompts; Motivation-based engagement prompts

SUMMARY:
Chemsex, the use of psychoactive drugs before or during sexual activity, is a growing public health concern associated with striking increases in HIV, particularly among men who have sex with men (MSM). This study proposes to optimize an app-based just-in-time adaptive intervention, called JomCare, which aims to reduce chemsex risk by delivering tailored support when a person is most likely to be vulnerable to chemsex risk behaviors and receptive to intervention, with the purpose of reducing risk and averting new HIV infections.

DETAILED DESCRIPTION:
Chemsex, the use of psychoactive drugs before or during sexual activity, is a growing public health concern due to its association with increased HIV transmission and other harms, particularly among men who have sex with men (MSM). Current estimates suggest that 9-26% of Malaysian MSM participate in chemsex, contributing to recent increases in HIV prevalence. In the absence of evidence-based interventions for chemsex, harm reduction strategies remain the most impactful approach to mitigating chemsex-associated harms. However, getting harm reduction interventions to MSM who engage in chemsex is a major challenge due to the spontaneous and dynamic nature of chemsex risk. Just-in-time adaptive interventions (JITAIs) delivered via smartphones represent a powerful strategy to deliver support by deploying tailored intervention when needed. Specifically, apps that incorporate JITAI can be more effective than traditional app-based interventions by addressing the dynamic nature of chemsex risk and capitalizing on users' changing states of vulnerability (heightened chemsex risk behaviors) and receptivity (willingness to engage in intervention), while also minimizing user burden, disruption, and habituation. Although JITAIs are increasingly being used in domains such as addiction, mental health disorders, physical inactivity, and obesity, research on JITAIs to address chemsex harm reduction is non-existent. In response, a smartphone app-based chemsex harm reduction JITAI called JomCare is developed that uses a machine learning algorithm to determine risk and deliver tailored support as needed. JomCare includes several 'pull' and 'push' intervention components based on the information-motivation-behavioral skills (IMB) model, and has demonstrated high feasibility and utility in our recent pilot work. However, little is known to guide which intervention components should be delivered in specific contexts to achieve maximum benefit, thus indicating the need to optimize JomCare. Framed by the multiphase optimization strategy (MOST) and building on our formative work, this study will optimize JomCare using a micro-randomized trial (MRT) to evaluate: i) which theory-driven intervention components are efficacious in reducing chemsex risk behaviors; and ii) which contexts influence the efficacy of JomCare. Specifically, this study will conduct a 90-day MRT of the JomCare JITAI among 482 chemsex-involved Malaysian MSM. Participants will be randomized twice daily via the app to receive: i) no prompt; ii) a generic engagement prompt; or iii) one of three IMB model-based engagement prompts. The specific aims of this application include: i) Evaluate the effects of any intervention (i.e., theory-driven or generic engagement prompts) versus no intervention on chemsex risk behaviors (proximal outcomes) at subsequent EMAs following randomization; ii) Compare the effects of theory-driven and generic engagement prompts on proximal outcomes; and iii) Examine contextual moderators of intervention on proximal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Cisgender man;
* HIV-negative or HIV status unknown;
* Having engaged in "chemsex" in the past 12 months (defined as using CAD, including crystal methamphetamine, mephedrone, GBL/GHB, and/or ecstasy/MDMA)
* Own a smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Enrolled in drug rehabilitation, substance use treatment, and narcotics or other behavioral intervention-based treatment
* Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender man
Enrollment: 482 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants engaged in chemsex risk behavior | Up to 6 months
  Use of chemsex-associated drugs, engagement in condomless anal sex, CAD overdose since the last EMA

CONTACTS AND LOCATIONS:
Overall Officials: Roman Shrestha, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shrestha R, Lim SH, Altice FL, Copenhaver M, Wickersham JA, Saifi R, Ab Halim MA, Naning H, Kamarulzaman A. Use of Smartphone to Seek Sexual Health Information Online Among Malaysian Men Who Have Sex with Men (MSM): Implications for mHealth Intervention to Increase HIV Testing and Reduce HIV Risks. J Community Health. 2020 Feb;45(1):10-19. doi: 10.1007/s10900-019-00713-x. PMID 31375976
- [Background] Rabbi M, Philyaw Kotov M, Cunningham R, Bonar EE, Nahum-Shani I, Klasnja P, Walton M, Murphy S. Toward Increasing Engagement in Substance Use Data Collection: Development of the Substance Abuse Research Assistant App and Protocol for a Microrandomized Trial Using Adolescents and Emerging Adults. JMIR Res Protoc. 2018 Jul 18;7(7):e166. doi: 10.2196/resprot.9850. PMID 30021714